CLINICAL TRIAL: NCT00933478
Title: A Trial of Clay Weight on the Ear Drum for Patulous Eustachian Tube
Status: Withdrawn | Type: Observational
Why Stopped: NSH REB has no record of this study being submitted for review
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: Clark Bartlett
Record Dates: First submitted 2009-07-06; First posted 2009-07-07 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2009-07

CONDITIONS: Patulous Eustachian Tube Dysfunction
Keywords: Patulous Eustachian Tube Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Patulous Eustachian Tube Dysfunction
  Interventions: Device: Clay

INTERVENTIONS:
Device: Clay — Small dime sized piece of clay.
  Other Names: Clay is used is Blue tac.

SUMMARY:
The Eustachian tube is a tube that connects the back of the nose with the ear. Its job is to keep the pressure on the inside of the eardrum close to the pressure outside the eardrum, so that the eardrum can vibrate properly. Usually this tube is closed, but it opens briefly during swallowing. In the condition called patulous eustachian tube, this tube is open all the time. This is a benign condition but it can be very bothersome to patients.

The incidence of patulous Eustachian tube dysfunction is about 0.3-6.6% of the population. However, about 15% of the people who have this condition are bothered enough by it that they seek medical attention. This condition is more common in females than males and is more common in adults than children.

Some of the common symptoms of patulous eustachian tube can include roaring tinnitus synchronous with nasal respiration, audible respiratory sounds, sensation of a plugged ear and fluctuating aural fullness.

In most cases the cause is idiopathic. Some predisposing factors include weight loss, stress,anxiety,fatigue, pregnancy, and temporomandibular joint syndrome. It can also be caused by adhesions in the nasopharynx following surgery on the adenoids. Sometimes it can be associated with medications such as diuretics and oral contraceptives. Neuromuscular disorders that cause atrophy such as multiple sclerosis, stroke and motor neuron disease have also been postulated to cause patulous eustachian tube.

The purpose of this trial is to learn more about the condition and help us learn about how the eardrum might be treated to prevent it vibrating with sounds or noises coming up the Eustachian tube.

The first part of the study will consist of a questionnaire to help to further define the symptoms of patulous eustachian tube, and to measure how severe these symptoms are.

Currently there are few treatments that are satisfactory for patients. Common surgical therapies include injections of various substances into the Eustachian tube opening including paraffin, Teflon,or gelfoam. Unfortunately, these methods are either temporary or have lead to serious complications including cerebral thrombosis and death (due to inadvertent injection into the carotid artery). Other treatments have focused on cauterizing the Eustachian tube opening but these have been either unsatisfactory or caused damage to the trigeminal nerve. Myringotomy and insertion of a ventilation tube has helped some patients but others have found that this increased the patient's discomfort.

The investigators have been treating patients recently by placing some putty like clay material on the eardrum, which stops it vibrating so much with the patient's own voice, and this appears to be quite effective for many patients. It is also easily removed if the patient does not find it helpful. However, the investigators do not really have a good idea of exactly which patients are helped by this, and which are not, and just how much their symptoms are helped, as well as how long the treatment helps them for.

DETAILED DESCRIPTION:
The Eustachian tube is a tube that connects the back of the nose with the ear. Its job is to keep the pressure on the inside of the eardrum close to the pressure outside the eardrum, so that the eardrum can vibrate properly. Usually this tube is closed, but it opens briefly during swallowing. In the condition called patulous eustachian tube, this tube is open all the time. This is a benign condition but it can be very bothersome to patients.1 The incidence of patulous Eustachian tube dysfunction is about 0.3-6.6% of the population. However, about 15% of the people who have this condition are bothered enough by it that they seek medical attention. This condition is more common in females than males and is more common in adults than children.1

Some of the common symptoms of patulous eustachian tube can include roaring tinnitus synchronous with nasal respiration, audible respiratory sounds, sensation of a plugged ear and fluctuating aural fullness.

In most cases the cause is idiopathic. Some predisposing factors include weight loss, stress,anxiety,fatigue, pregnancy, and temporomandibular joint syndrome. It can also be caused by adhesions in the nasopharynx following surgery on the adenoids. Sometimes it can be associated with medications such as diuretics and oral contraceptives. Neuromuscular disorders that cause atrophy such as multiple sclerosis, stroke and motor neuron disease have also been postulated to cause patulous eustachian tube.1 -2

The purpose of this trial is to learn more about the condition and help us learn about how the eardrum might be treated to prevent it vibrating with sounds or noises coming up the Eustachian tube.

The first part of the study will consist of a questionnaire to help to further define the symptoms of patulous eustachian tube, and to measure how severe these symptoms are.

Currently there are few treatments that are satisfactory for patients. Common surgical therapies include injections of various substances into the Eustachian tube opening including paraffin, Teflon,or gelfoam. Unfortunately, these methods are either temporary or have lead to serious complications including cerebral thrombosis and death (due to inadvertent injection into the carotid artery). Other treatments have focused on cauterizing the Eustachian tube opening but these have been either unsatisfactory or caused damage to the trigeminal nerve. Myringotomy and insertion of a ventilation tube has helped some patients but others have found that this increased the patient's discomfort.3-4

We have been treating patients recently by placing some putty like clay material on the eardrum, which stops it vibrating so much with the patient's own voice, and this appears to be quite effective for many patients. It is also easily removed if the patient does not find it helpful. However, we do not really have a good idea of exactly which patients are helped by this, and which are not, and just how much their symptoms are helped, as well as how long the treatment helps them for.

We have not found any permanent hearing loss from putting the putty on the eardrum.

Subject Selection:

There will be approximately twenty patients in total. The absolute number will depend on the number of patients that present with patulous eustachian tube and agree to participate. All patients will have been referred to our clinic from other otolaryngologists for treatment of this particular problem. These patients will be selected if they meet the diagnostic criteria for patulous eustachian tube. There will be no exclusion criteria based on age or gender.

Research Plan There will be no randomization procedure, as all patients will receive treatment for their condition. The investigators will not be blinded, as they are the only ones able to perform the treatment.

The patients will be asked to follow up in clinic as per his regular visit protocol. They are usually booked for four-month follow up appointments. If they have concerns they will be asked to call and book an appointment for an earlier date.

There will be no laboratory testing. The amount of clay to be used is the amount to cover the size of a dime. If there are any concerns or adverse reactions to treatment the patient will have the treatment stopped. The clay or steristrip will be removed.

Analysis of Data The data will be compiled and sent to a member of the statistics department at Dalhousie University. All identifying data will be removed. The pre-treatment values will then be compared to post treatment values to see if a statistical significance exists.

Confidentiality All data will kept in a locked filing cabinet and office for 25 years, and only research staff will have access to it. The data will be analyzed using various computer programs, such as Gaitview 2002, Microsoft Office programs, and SPSS for statistical analysis. The data on these programs will only be available to research staff via a secure password. Names of patients will only be available to research staff, and numerical codes will be used in any presentations or publications of the data. The research team will collect and use only the information they need to judge the safety and usefulness of the study. This information will only be used for the purposes of this study.

Only Dr.Bance and Dr.Bartlett will have access to the study data.

Harms There are very few risks to this trial. It is generally a well-tolerated procedure. The biggest risk is failure of the procedure. It does not work for everyone.

The laser measurements of the eardrum are without risk. This laser does not damage tissue.

Putting the steri-strip or clay weight on the eardrum may carry about a 1 in 300 risk of a small puncture to the eardrum. Of these, over 95% heal up by themselves, but some may need to be repaired. This, however, is currently our preferred first line treatment for patulous Eustachian tube currently anyway.

Benefits

There is no financial incentive to join the trial. The major benefit will be a potential resolution of the symptoms of patulous eustachian tube.

The societal benefits are an easy safe treatment for this condition.

Financial Compensation

There is no financial compensation for anyone involved in this trial. This includes participants and researchers.

ELIGIBILITY:
Inclusion Criteria:

* presence of condition (patulous eustachian tube dysfunction)

Exclusion Criteria:

* Hole in Tympanic Membrane.
* Allergy to Blue tac

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected if they meet the diagnostic criteria for patulous eustachian tube.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07 (Estimated); Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Amount recorded improvement with treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clark G Bartlett, MD, Principal Investigator — Dalhousie Department of Otolaryngology
Locations (1):
- Victoria General Hospital, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] O'Connor AF, Shea JJ. Autophony and the patulous eustachian tube. Laryngoscope. 1981 Sep;91(9 Pt 1):1427-35. doi: 10.1288/00005537-198109000-00003. PMID 7346684
- [Background] Virtanen H, Palva T. Surgical treatment of patulous eustachian tube. Arch Otolaryngol. 1982 Nov;108(11):735-9. doi: 10.1001/archotol.1982.00790590057016. PMID 7138369
- [Background] Sehhati-Chafai-Leuwer S, Wenzel S, Bschorer R, Seedorf H, Kucinski T, Maier H, Leuwer R. Pathophysiology of the Eustachian tube--relevant new aspects for the head and neck surgeon. J Craniomaxillofac Surg. 2006 Sep;34(6):351-4. doi: 10.1016/j.jcms.2006.03.006. Epub 2006 Jul 21. PMID 16859910
- [Result] Cairns W. The patulous Eustachian tube syndrome. Palliat Med. 1998 Jan;12(1):59-60. doi: 10.1191/026921698671963177. No abstract available. PMID 9616461